CLINICAL TRIAL: NCT05342233
Title: Comparison of Conservative and Endovascular Treatment for Spontaneously Isolated Superior Mesenteric Artery Dissection: A Real-world, Multicenter, Observational Study
Brief Title: Comparison of Conservative and Endovascular Treatment for Spontaneously Isolated Superior Mesenteric Artery Dissection
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: The First Medical Center of Chinese PLA General Hospital (Other); West China Hospital (Other); Renmin Hospital of Wuhan University (Other); Peking University Shenzhen Hospital (Other); Affiliated Hospital of Chengde Medical University (Other); Second Affiliated Hospital of Nanchang University (Other); Henan Provincial People's Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Principal Investigator, xueguanwaike, Professor, Xiangya Hospital of Central South University
Other Study IDs: ISMAD2022
Record Dates: First submitted 2022-04-10; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Spontaneous Isolated Superior Mesenteric Artery Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular treatment Group: Patients receiving endovascular treatments
- Conservative treatment Group: Patients receiving conservative treatments, including blood pressure control, bowel rest, antithrombotic therapy, nutrition treatment and pain management.

SUMMARY:
Spontaneous isolated superior mesenteric artery dissection(SISMAD) is an increasingly diagnosed disease. However, prospective, multicenter studies that can provide evidence to support clinical decisions are very limited. This study aims to compare the therapeutic efficacy of conservative and endovascular treatment for SISMAD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and above;
2. Isolated superior mesenteric artery dissection with clear symptoms or history and confirmed by CTA
3. Signed informed consent forms, willing to receive treatments

Exclusion Criteria:

1. Symptoms are severe and patients need exploratory laparotomy;
2. Patients with aortic dissection, iliac artery dissection, or autoimmune vasculitis;
3. Patients with mental illness cannot cooperate subjectively;
4. Patients who are allergic to contrast agents, or contraindicated to conservative treatment drugs, and cannot be treated with drugs;
5. Pregnancy and breastfeeding women, or patients who have recent birth plans;
6. Patients who are participating in other clinical projects;
7. Patients are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms or history of isolated superior mesenteric artery dissection and confirmed by CTA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 5 years
  Mortality during follow-up period
Rate of symptom relief | up to 5 years
  Rate of symptom relief during follow-up period

SECONDARY OUTCOMES:
Reintervention rate | Follow-up period（ 5 years）
  Reintervention related to SISMAD after treatments during follow-up period
Recurrence rate | Follow-up period（5 years）
  SISMAD Recurrence after treatments during follow-up period
Disease-related complications | Follow-up period（5 years）
  Disease-related complications after treatments during follow-up period
Complete remodeling rate of superior mesenteric artery dissection | Follow-up period（5 years）
  Complete remodeling rate of superior mesenteric artery dissection after receiving different treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China